CLINICAL TRIAL: NCT01703494
Title: Fecal Microbiota Transplantation for Relapsing Clostridium Difficile Infection
Brief Title: Fecal Transplant for Relapsing C. Difficile Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Colleen Kelly (Other)
Responsible Party: Sponsor-Investigator, Colleen Kelly, Clinical Assistant Professor of Medicine, The Miriam Hospital
Organization: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21DK093839-01A1 (NIH)
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Clostridium Difficile
Keywords: C. difficile; fecal transplant; stool transplant; fecal flora reconstitution; fecal microbiota transplant; FMT
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal Microbiota Transplantation (Active Comparator): After completing at least a 10 day course of vancomycin for treatment of the most recent acute C. difficile infection, subjects will receive fecal Microbiota Transplant (FMT) with a 300 mL donor fecal suspension delivered via colonoscopy.
  Interventions: Biological: Fecal Microbiota Transplantation
- Sham Fecal Microbiota Transplantation (Sham Comparator): After completing at least a 10 day course of vancomycin for treatment of the most recent acute severe C. difficile infection, subjects will receive a 300 mL infusion of a sham (autotransfusion) fecal solution at colonoscopy.
  Interventions: Biological: Sham Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Fecal microbiota transplantation (FMT) involves administering fecal material from a healthy individual (donor) to a sick patient (with relapsing C. difficile infection) to restore missing components of normal intestinal flora. After completing at least a 10 day course of vancomycin for treatment of the most recent acute C. difficile infection, subjects will receive fecal microbiota transplantation (FMT) with a 300 mL donor fecal suspension delivered via colonoscopy.
  Other Names: FMT; fecal bacteriotherapy; fecal flora reconstitution; stool transplant
  Arms: Fecal Microbiota Transplantation
Biological: Sham Fecal Microbiota Transplantation — After completing at least a 10 day course of vancomycin for treatment of the most recent acute C. difficile infection, subjects will receive a sham fecal microbiota transplantation (FMT) with a 300 mL sham fecal suspension delivered via colonoscopy. This sham solution will be a reinfusion of the subject's own stool.
  Arms: Sham Fecal Microbiota Transplantation

SUMMARY:
There has been an alarming increase in the incidence and severity of Clostridium difficile infection (CDI) in North America over the past decade. Relapsing infection is a common problem in patients treated for CDI, often requiring prolonged and expensive courses of oral vancomycin with limited alternative treatment options. This study will determine if fecal microbiota transplantation, which involves administering fecal flora from a healthy stool donor to a patient with relapsing CDI, is an effective and safe treatment.

DETAILED DESCRIPTION:
Clostridium difficile is an increasingly common infection. The number of hospital discharges for which C. difficile was listed as the first diagnosis more than doubled between 2000 and 2003. In addition to occurring more frequently, there is an epidemic of serious cases which are more refractory to therapy and which have high rates of colectomy and death. Most commonly, C. difficile infection (CDI) is associated with use of antimicrobial agents that are thought to alter the normal bacterial flora of the gastrointestinal tract so as to permit colonization and/or proliferation and toxin elaboration by C. difficile. Though the precise mechanisms by which this occurs are still incompletely understood, depletion of physiologic microflora, in particular Bacteroides species may play an important role. Most patients with CDI respond to a course of oral metronidazole or vancomycin, however, up to 20% of patients relapse after initial treatment. Current guidelines recommend a tapering course of vancomycin after a second recurrence, however up to 60% of patients still do not respond to this treatment strategy or develop further recurrence after the vancomycin is stopped. Use of antimicrobials to treat CDI may predispose these patients to further relapses through the maintenance of disturbed intestinal flora and may contribute to the emerging problem of drug resistance.

"Fecal Microbiota Transplantation" (FMT) is a novel treatment approach which involves administration of feces from a healthy (donor) individual into a patient with relapsing CDI to promote recolonization with missing components of normal intestinal flora. Numerous case reports and retrospective case series have suggested benefit of FMT in patients with severe or recurrent CDI with cure rates as high as 100% and a mean cure rate of 89% for the nearly 300 cases reported in the world literature. Although efficacy has been documented in these case reports, to date there has not been a published prospective clinical trial of FMT for CDI.

The proposed study would be the first randomized, double-blind, placebo (sham) controlled clinical trial to determine whether FMT delivered at colonoscopy is effective at preventing further relapse in patients who have suffered from at least a 3rd recurrence of CDI despite receiving standard treatment. The investigators hypothesize that FMT is superior to placebo in preventing relapse after treatment of CDI with vancomycin. As a result of this study, the investigators will have preliminary efficacy data for this novel treatment approach for recurrent CDI. The investigators will be better prepared to test the efficacy of FMT in future multicenter clinical trials. This research will advance clinical care, potentially impacting the protocol for treatment of relapsing C. difficile infection worldwide. This proposal includes collaboration with an investigator capable of performing microbiome analyses on specimens collected as part of the trial and will further understanding of the intestinal microflora in health and disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatients (age ≥18 and <75) referred to one of the study centers after suffering a third (or further) documented episode CDI and
2. who have failed to maintain CDI cure after standard therapy with oral vancomycin.

   * Previous treatment with at least one course of tapered/pulse dose vancomycin as per SHEA-IDSA C difficile treatment guidelines or -Inability to taper or stop vancomycin without developing diarrhea requiring anti-infective therapy. -

Exclusion Criteria:

* Patients who are aged 75 years or greater.
* Patients who are pregnant
* Patients who are nursing
* Patients who are incarcerated
* Patients with cognitive impairment or severe neuropsychiatric co morbidities who are incapable of giving their own informed consent
* Patients who are immunocompromised specifically:
* HIV infection (any CD4 count)
* AIDS-defining diagnosis or CD4<200/mm3
* Inherited/primary immune disorders
* Immunodeficient or Immunosuppressed due to medical condition/medication:
* Current or recent (<3 most) treatment with anti-neoplastic agent
* Current or recent (<3 mos) treatment with any immunosuppressant medications (including but not limited to monoclonal antibodies to B and T cells, anti-TNF agents, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine), calcineurin inhibitors (tacrolimus, cyclosporine), mycophenolate mofetil). Subjects who are otherwise immunocompetent and have discontinued any immunosuppressant medications 3 or more months prior to enrollment may be eligible to enroll.
* Patients with a history of severe (anaphylactic) food allergy
* Patients who have previously undergone FMT
* Patients who are unwilling or unable to undergo colonoscopy
* Patients with untreated, in-situ colorectal cancer
* Patients with a history of inflammatory bowel disease (ulcerative colitis, Crohn"s disease or microscopic colitis) or irritable bowel syndrome
* Unable to comply with protocol requirements
* Patients who are American Society of Anesthesiologists (ASA) Physical Status classification IV and V
* Patients with acute illness or fever on the day of planned FMT will be excluded (not undergo randomization or treatment with FMT) with the option of including that subject at a future date.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Cure | 8 weeks
  Resolution of diarrhea (i.e., fewer than three unformed stools for two consecutive days), with maintenance of resolution for the duration of the 8 week follow-up period and no further requirements for anti-infective therapy for C. difficile infection). Subjects who meet this definition will be considered cured regardless of results of follow-up stool testing for C. difficile.

SECONDARY OUTCOMES:
Clinical Failure | 8 weeks
  Persistence or development of diarrhea and the need for additional anti-infective therapy for C. difficile infection with or without positive stool testing (PCR) for C. difficile. Upon clinical failure, subject's treatment will be unblinded and those who received sham Fecal Microbiotia Transplantation (FMT) may chose to receive open label FMT using donor stool. Subjects, who received true FMT and develop clinical failure, may chose to undergo a second FMT using an alternate donor.

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months
  Subjects will be followed closely for significant adverse events and adverse events during the 8 week follow up period post-FMT and the development of new medical conditions/diagnoses or changes in medical conditions/medications will be determined at 6 month follow up contact. Adverse events will be tabulated by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen R Kelly, MD, Principal Investigator — Lifespan/ The Miriam Hospital; Lawrence J Brandt, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Montefiore Medical Center, The Bronx, New York
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Khoruts A, Dicksved J, Jansson JK, Sadowsky MJ. Changes in the composition of the human fecal microbiome after bacteriotherapy for recurrent Clostridium difficile-associated diarrhea. J Clin Gastroenterol. 2010 May-Jun;44(5):354-60. doi: 10.1097/MCG.0b013e3181c87e02. PMID 20048681
- [Background] Persky SE, Brandt LJ. Treatment of recurrent Clostridium difficile-associated diarrhea by administration of donated stool directly through a colonoscope. Am J Gastroenterol. 2000 Nov;95(11):3283-5. doi: 10.1111/j.1572-0241.2000.03302.x. No abstract available. PMID 11095355
- [Background] Yoon SS, Brandt LJ. Treatment of refractory/recurrent C. difficile-associated disease by donated stool transplanted via colonoscopy: a case series of 12 patients. J Clin Gastroenterol. 2010 Sep;44(8):562-6. doi: 10.1097/MCG.0b013e3181dac035. PMID 20463588
- [Background] Kelly CR, de Leon L, Jasutkar N. Fecal microbiota transplantation for relapsing Clostridium difficile infection in 26 patients: methodology and results. J Clin Gastroenterol. 2012 Feb;46(2):145-9. doi: 10.1097/MCG.0b013e318234570b. PMID 22157239
- [Derived] Kelly CR, Khoruts A, Staley C, Sadowsky MJ, Abd M, Alani M, Bakow B, Curran P, McKenney J, Tisch A, Reinert SE, Machan JT, Brandt LJ. Effect of Fecal Microbiota Transplantation on Recurrence in Multiply Recurrent Clostridium difficile Infection: A Randomized Trial. Ann Intern Med. 2016 Nov 1;165(9):609-616. doi: 10.7326/M16-0271. Epub 2016 Aug 23. PMID 27547925